CLINICAL TRIAL: NCT05023447
Title: The BRIDGE Project: A Feasibility Randomised Controlled Trial of Brief, Intensive Assessment and Integrated Formulation for Young People (Age 14-24) Early in the Course of Borderline Personality Disorder
Brief Title: The BRIDGE Project
Acronym: BRIDGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GN21MH147
Record Dates: First submitted 2021-07-09; First posted 2021-08-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDGE Intervention (+Service as Usual) (Experimental): Brief, intensive assessment and integrated formulation (BRIDGE) intervention is guided by the evidence base of Cognitive Analytic Therapy (CAT) with young people (aged 14-25) with features of BPD using an early intervention model and in collaboration with an established Glasgow programme, Intensive Support and Monitoring Service (ISMS). ISMS focuses on reaching a shared formulation with the young person and the multi-agency system that supports them.
  BRIDGE is delivered over 3-6 months and includes :- an intensive assessment, including BPD symptoms, copresenting difficulties, neurodevelopmental profile, life events history and psychosocial functioning; up to 16 sessions of Cognitive Analytic Therapy (CAT) and the development of a shared formulation with a multi-agency group. Further development of this formulation with the young person, using CAT principles (Reformulation, Recognition and Revision) and, where clinically applicable, their family and service-providers.
  Interventions: Behavioral: BRIDGE Intervention; Behavioral: Service as Usual
- Service as Usual (Active Comparator): Services as Usual (SAU) For participants randomised to SAU, a routine letter of their participation will be shared with their service provider(s), including their GP. SAU, is likely to range from social services, mental-health services, forensic services to no services in some cases. Pathways to care and service involvement will be mapped and described for each participant. Treatment fidelity to SAU will therefore not be assessed, but the nature and intensity of SAU in different contexts will be described in detail through the qualitative process evaluation.
  Interventions: Behavioral: Service as Usual

INTERVENTIONS:
Behavioral: BRIDGE Intervention — Intensive clinical assessment; >16 sessions of Cognitive Analytic Therapy (CAT); Development of a shared formulation
  Arms: BRIDGE Intervention (+Service as Usual)
Behavioral: Service as Usual — Likely to range from social services, mental-health services, forensic services to no intervention

SUMMARY:
The BRIDGE project: A feasibility randomised controlled trial of brief, intensive assessment and integrated formulation for young people (age 14-24) early in the course of borderline personality disorder.

DETAILED DESCRIPTION:
This project is the first step in testing a new intervention programme, called BRIDGE (Brief, Intensive Assessment and Integrated Formulation), for young people early in the course of Borderline Personality Disorder (BPD). The BRIDGE Project will help us find out whether we can do a much bigger study in the future that will tell us whether BRIDGE works well. BPD is characterised by long standing difficulty in managing emotional responses, personal relationships, impulse control and self-image. Research shows that individuals with BPD may experience discrimination and resulting stigmatisation by both the public and health care professionals. Many adolescents and young people with complex needs and high suicide risk are left under-diagnosed and untreated. As a result, young people with BPD are frequently not in education or training and experience challenging relationships with friends and families. The overall aim of the study is to assess the possibility of providing a treatment programme for young people with BPD symptoms in the general population, who may or may not be accessing any mental health services. First, we need to see whether young people are comfortable with random allocation to BRIDGE (AND service as usual) or Service-as-usual (ALONE) (a bit like tossing a coin). Second, we need to find out whether enough young people want to be involved. Third, whether we can find out the information we need about them and can follow up enough young people later. The proposed study will try to find these things out, so that we can design a future, bigger, study to find out whether BRIDGE is good value for young people with BPD.

ELIGIBILITY:
Inclusion Criteria:

* Cut off score of 11 out of 15 on the self-reported SCID-II BPD questionnaire AND subthreshold (3 or 4 out of 9 domains) or threshold (5 and above out of 9 domains) criteria on the SCID-II DSM-V (BPD Module)
* Age 14-25

Exclusion Criteria:

* Currently receiving psychological/counselling /psychotherapeutic treatment for BPD
* Has received psychological/counselling/psychotherapeutic intervention for over 8 sessions in the last 3 months
* Severe or profound intellectual disability, that would preclude full engagement in talking therapy
* Receiving Intensive psychiatric treatment at the time of study entry, for conditions such as acute psychosis or severe eating disorder
* Non-English speaking

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment & Retention rates | Continuous over 3 year study period
  The number of participants recruited for randomisation and the number retained to follow-up (12 & 24wks post randomisation).

SECONDARY OUTCOMES:
Acceptability of trial processes and interventions | Continuous over 3 year study period
  Explored through qualitative interviews
Process Evaluation | Continuous over 3 year study period
  Theory of change and logic modelling will be explored to capture the process behind intervention effects.

OTHER OUTCOMES:
Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II) PQ-BPD | Screening; Pre-randomisation
  15 Item Questionnaire for Borderline Personality Disorder
Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II) DSM-V | Screening/Pre-randomisation
  Clinical interview using the SCID-II DSM-V
KIDSCREEN-10 Index | Screening/Pre-randomisation
  Health Questionnaire for Children and Young People
KIDDIE Schedule for Affective Disorders and Schizophrenia Present and Lifetime Version (K-SADS-PL) | within 2 weeks of randomisation (baseline)
  Questionnaire for affective disorders and schizophrenia
Adverse Childhood Experiences Scale | within 2 weeks of randomisation (baseline)
  Questionnaire for Adverse Childhood Experiences
The Autism Symptom Self Report for Adolescents (ASSERT) Scale | within 2 weeks of randomisation (baseline)
  Questionnaire for symptoms of Autism
Adult ADHD Self-Report Scale (ASRS) | within 2 weeks of randomisation (baseline)
  Questionnaire for ADHD symptoms in adulthood
Borderline Symptoms List (BSL) | Baseline and Follow-up (12 and 24weeks post randomisation)
  Questionnaire for symptoms of Borderline Personality Disorder (BPD)
Sheehan's Disability Scale (SDS) | Baseline and Follow-up (12 and 24weeks post randomisation)
  Assessment of functional impairment
Difficulties in Emotional Regulation Scale-Short Form (DERS-SF) | Baseline and Follow-up (12 and 24weeks post randomisation)
  Questionnaire to assess emotion regulation
Patient Health Questionnaire-9 (PHQ-9) | Baseline and Follow-up (12 and 24weeks post randomisation)
  General health questionnaire
EuroQol-5D-5L (EQ-5D-5L) | Baseline and Follow-up (12 and 24weeks post randomisation)
  Quality of Life questionnaire
Suicidal Ideation Scale | Baseline and Follow-up (12 and 24weeks post randomisation)
  Questionnaire for suicidal ideation
Vocational and Educational Functioning | Baseline and Follow-up (12 and 24weeks post randomisation)
  Measure of functioning in domains of work and education

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika Gajwani, Dr, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde Clinical Research and Development Central Office, Paisley, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The PI will manage access rights to the data set. We anticipate that anonymised trial data may be shared with other researchers to contribute to the emerging BPD evidence base.

REFERENCES:
- [Derived] Gajwani R, Sim F, McAllister K, Smith H, McIntosh E, Moran P, Ougrin D, Smith M, Gumley AI, Chanen AM, Minnis H. The BRIDGE project: a feasibility randomised controlled trial of brief, intensive assessment and integrated formulation for young people (age 14-24) with features of borderline personality disorder (Protocol). Front Psychiatry. 2024 Sep 24;15:1389578. doi: 10.3389/fpsyt.2024.1389578. eCollection 2024. PMID 39381608

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT05023447/Prot_SAP_000.pdf